CLINICAL TRIAL: NCT00813631
Title: The Effect on an Ionic Silver Dressing in Head and Neck Patients With Malignant Fungating Wound
Acronym: MFW
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: We-Yu Hu, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200804050R
Record Dates: First submitted 2008-12-21; First posted 2008-12-23 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-03

CONDITIONS: Head and Neck Neoplasms; Head and Neck Cancer; Wounds; Ulcer
Keywords: Malignant fungating wound; Head and neck; Ionic silver-releasing dressing; Wound care; RCT
MeSH Terms: conditions — Head and Neck Neoplasms; Wounds and Injuries; Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- silver-releasing dressings (Experimental): Silver, in its common ionic (active) form (Ag+), is particularly attractive as an antibacterial agent because it can be readily incorporated into dressing materials. Silver-dressing are wound products designed to control infection and provide a wound environment conducive to management exudates, pain, and malodour.
  Interventions: Other: silver-releasing dressings

INTERVENTIONS:
Other: silver-releasing dressings — Experimental group are accepted primary dressing the AQUACEL Ag. control group are provided with the AQUACEL on the wound surface. Wound specialist or primary nurses undertaking wound care are informed by inclusion criteria that the treatment shall be adhered to during the two-week study period.All wounds are cleansed with sterile saline prior to assessment and dressing application.The sterile, non-woven sodium carboxymethylcellulose primary AQUACEL Ag with 1.2% ionic silver.Each secondary dressing is covered a sterile gauze.Dressings are changed between daily assessments when judged necessary.Patients attended the wound ward weekly for treatment evaluation. All participating clinics used the same wound management guidelines and data collection forms.
  Other Names: AqCel Ag,AQUACEL,AQUACEL Ag,Aq Cel

SUMMARY:
Background. Malignant fungating wounds(MFW) are caused by cancerous cells invading skin tissue, which exhibit increased bacterial burdens that not only result in a negative physical impact (odour, exudates, pain, and infection) on patients, impairing their quality of life, but they also increase treatment costs. A systematic review of the effectiveness of that the silver-releasing dressing in the management of infected chronic wounds can help enhance control of wound bed infection and inflammation, tissue management, moisture balance, and protect wound edge. However, few studies have examined the effects on people with MFW.

Hypothses In this study that the hypothesized that cancer patients in the ionic silver dressing group will perception higher quality of life compared to patients in the control group who receive non-ionic silver dressing. In addition, we hypothesized that cancer patients who also receive ionic silver dressing will have lower level of symptom distress at end of study compared to patients in the control group receive non-ionic silver dressing care.

DETAILED DESCRIPTION:
Introduction. At the beginning of the 21st century, cancer is increasing in the aging population and patients often have a greater life expectancy than they did 40 years ago (Payne et al 2004). As people age, and the incidence of cancer increases, it is essential to push the frontiers of oncology care to meet the symptom management needs of these patients. For many, cancer has become a slowly progressive, chronic disease - a change that brings with it particular challenges for oncology nurses (Hoskin and Makin 1998). A systematic review of the effectiveness of that the silver-releasing dressing in the management of infected chronic wounds can help enhance control of wound bed infection and inflammation, tissue management, moisture balance, and protect wound edge. This study is designed to assess the effects of ionic silver dressing (AQUACEL Ag) in head and neck patients with malignant fungating wound (MFW) on the quality of life, symptom distress and wound bed changed of patients with MFW

Definition of MFW. Malignant Fungating wounds arise as a result of infiltration of the structures of the skin by malignant cells. These cells may arise from primary skin cancer, an underlying malignant tumor or through metastasis spread from a distant malignant tumor(Punder, 1998).A fungating cancer is a primary or secondary malignant growth in the skin which has ulcerated and results in pain, exudates, bleeding, infection and malodour(Twycross, 1995) .A malignant tumor will invade and destroy adjacent tissues and can spread to other tissues with in cells that break off and travel in the blood or lymph system. It can develop its own blood supply, sometime outgrowing it and causing the tumor to become necrotic in the middle(Mera, 1997).Dealey(1994) states that, as the tumor extends, capillaries rupture, leading to epithelium results in ulceration through the skin, and lesions presents as a fungating, foul-smelling mass(Daeley, 1994).Fungating malignant wounds are caused by the infiltration of the skin and its supporting blood and lymph vessels by a local tumor or as a result of metastasis growth from the primary tumor. Unless the malignant cells are checked by single or combination cancer treatments the fungation extends with the potential for causing massive damage at the wound site through a combination of proliferate growth, loss of vascularity and ulceration(Mortimer, 1998) .A fungating wound is defined as a cancerous lesion involving the skin, which is open and may be draining. The lesion may be result of a primary cancer or metastasis to the skin from a local tumor or from a tumor in a distant site. It may take the form of a cavity, an open area on the surface of the skin, skin nodules, or a nodular growth extending from the surface of the skin(British Columbia Cancer Agency, 2001) .As the malignant cells multiply in the skin they form a tumour that enlarges causing disruption of skin capillaries and lymph vessels, eventually leading to tissues Hypoxia and subsequent skin necrosis.

Infection control of MFW. All chronic wounds contain bacteria. Kingsley(2003) state that the change in numbers of bacteria and the body's response as a continuum, rating from contamination to infection(Kingsley, 2003). Contamination is mean that the bacteria present on the wound surface but are not proliferating and have no clinic effect; colonised imply bacteria have proliferated, but there is no host reaction; critical colonisation occurs where the body's local host response starts to be initiated, but there are no systemic sign of infection; Infection is point in time when the bacteria have multiplying and invaded deeper tissues, healing is impaired and produced a systemic host reaction(Jacqui. Fletcher, 2005; Verdu Soriano , Rueda Lopez, Martinez Cuervo, & Soldevilla Agreda 2004) .

Clinical recognition of these rating stages is not easy because there are no clear descriptors. However, Soriano et al (2004) defined classification according to the number of bacteria present in the wound bed: Contamination-≦103 colony-forming unit (CFUs) per gram of tissues; colonised -≦104 CFUs ; Infection -≧105 CFUs. Cutting and White noted several aspects of wound infection such as: serous drainage with concurrent inflammation, discoloured granulation tissue, pocketing at the wound base, unexpected pain , foul odour, increase in exudates, exudates that becomes purulent instead of serous, and wound breakdown(White & Cutting, 2006).

In the MFW, the presence of hypoxic necrotic tissues within the wound provides an excellent medium for growth of aerobic and anaerobic bacteria(J. Clark, 2002). Anaerobic and aerobic bacteria thrive in these conditions, giving rise to excessive malodour wound exudates(Haisfield-Wolfe & Rund 1997). Lo et al (2006) survey of seventy cancer patients with MFW in Taiwan, the study found that the 60.3% wound bed presented necrotic tissue ; malodour was present in 50% of patients ; 81.4% shows moderate to large exudates and 71.4% reported purulent(Lo, 2006). According above the data, infection has emerged as a major health problem during the patient suffers MFW.

Ionic silver dressing. Silver, in its common ionic (active) form (Ag+), is particularly attractive as an antibacterial agent because it can be readily incorporated into dressing materials. When the materials contact an aqueous environment, the silver complex contained in them is dissociated (Ovington 2004, White & Cutting 2006). The mechanism of action for Ag+ is that it binds to bacterial cell DNA, and enzymes, and proteins in the cell wall. Once the silver cation attaches to these sites, it alters their structure, resulting in structural and functional changes in the bacterial cell (Ovington 2004).It is suggested by numerous authors that silver dressings should be utilized when critical colonization within a wound occurs (Ovington 2004, White & Cutting 2006, Lo et al 2008). Therefore, this study research questions is (1)What are the effects of ionic silver dressing (AQUACEL Ag)in head and neck patients with malignant fungating wound, as compared to hydrofiber dressing(AQUACEL), on the individual perception subjective quality of life?(2) What are the effects of ionic silver dressing (AQUACEL Ag) in head and neck patients with malignant fungating wound, as compared to hydrofiber dressing (AQUACEL) alone, on the symptom distress and wound bed changed of patients receiving ionic silver dressing (AQUACEL Ag) for cancer patients?

ELIGIBILITY:
Inclusion Criteria:

* (1.)Had a first time diagnosis of cancer of the breast or head and neck with MFW;
* (2)Are at least more than 18 years of age or older, in order to focus the study on an adult population
* (3)Present at malignant fungating wound more than one month old;
* (4)Are able to speak and understand Chinese, in order to understand the consent form and the intervention and complete the study questionnaires

Exclusion Criteria:

* (1) patients conscious unclear;
* (2) Had seriously medical or psychology, such as hemodialysis;
* (3) Had other comorbidity may interfere with intervention ion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
The data are collected using questionnaires completed by the subjects themselves.In this study , the primary outcome is health-related quality of life (HRQOL) | Each group was followed up for two week

SECONDARY OUTCOMES:
Also, the Secondary outcome measure using the modified Schulz Malignant Wound Assessment Tool (mSMWAT) | Each group was followed up for two week

CONTACTS AND LOCATIONS:
Overall Officials: We-Yu Hu, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan